CLINICAL TRIAL: NCT04258501
Title: An Exploratory Study of Efficacy and Tolerance on Selected Natural Extracts, With the Potential of Reducing Post Prandial Blood Glucose Response, in Healthy Indian Adult Subjects
Brief Title: Exploratory Study of Efficacy on Selected Natural Extracts Reducing Post Prandial Blood Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Lambda Therapeutic Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FDS-NAA-0334
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Blood Glucose
MeSH Terms: interventions — Morus alba; elderberry extract; Curcumin

STUDY DESIGN:
Intervention Model Description: Randomized, balanced, incomplete block design exploratory study of efficacy, with 8 active treatments (4 treatments per subject; 35 or 37 subjects per treatment) compared to a reference treatment (all 72 subjects).
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was generated by the bio-statistician CRO. Subjects and key study team personnel were blinded as much as possible with regard to the identification of specific treatments but their distinctive colors, flavors or tastes could not be masked.
  To ensure the study team was not apparently aware of the treatments being administered to subjects, persons who were involved in the preparation of test products were not involved in rest of the study.
  The sponsors team was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Mulberry fruit extract (Experimental): 1.5 g of mulberry fruit powdered extract mixed into a bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Mulberry fruit
- Mulberry leaf extract (Experimental): 1.0 g of mulberry leaf powdered extract mixed into aa bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Mulberry leaf
- White bean extract (Experimental): 3 g of white bean powdered extract mixed into a bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: White bean
- Apple extract (Experimental): 2 g of apple powdered extract standardized in phloridzin mixed into a bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Apple
- Elderberry extract (Experimental): 2 g of elderberry powder extract mixed into a bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Elderberry
- Turmeric extract (Experimental): 0.18 g of curcumin powdered extract mixed into a bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Turmeric
- Turmeric extract + Apple extract (Experimental): 0.18 g of curcumin powdered extract + 2 g of apple powdered extract standardized in phloridzin mixed into a bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Apple; Other: Turmeric
- Turmeric extract + Elderberry extract (Experimental): 0.18 g of curcumin powdered extract + 2 g of elderberry powder extract mixed into aa bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Elderberry; Other: Turmeric
- Rice porridge control (Placebo Comparator): Bowl containing 60 g of extruded rice + 300 ml of boiling water
  Interventions: Other: Rice porridge

INTERVENTIONS:
Other: Mulberry fruit
  Arms: Mulberry fruit extract
Other: Mulberry leaf
  Arms: Mulberry leaf extract
Other: White bean
  Arms: White bean extract
Other: Apple
  Arms: Apple extract; Turmeric extract + Apple extract
Other: Elderberry
  Arms: Elderberry extract; Turmeric extract + Elderberry extract
Other: Turmeric
  Arms: Turmeric extract; Turmeric extract + Apple extract; Turmeric extract + Elderberry extract
Other: Rice porridge
  Arms: Rice porridge control

SUMMARY:
Randomized, balanced, incomplete block design exploratory study of efficacy, with 8 active treatments (4 treatments per subject; 35 or 37 subjects per treatment) compared to a reference treatment (all 72 subjects).

DETAILED DESCRIPTION:
Incomplete block design cross over study in which the subjects consumed commercial rice porridge (60 grams of extruded rice to which 300 ml of boiling water was added) in the morning in a fasted state. On each visit one of the seven different natural exacts was mixed into this porridge just before consumption. The reference was consumed by all subjects and consisted of plain porridge with no extract added.

ELIGIBILITY:
Inclusion Criteria:

1. Is the volunteer willing to give his consent to participate in the study in writing?
2. Is the volunteer between the age of >20 and <50 yrs?
3. Is the volunteer's Body Mass Index (BMI) in between >18 and <25 kg/m2?
4. Lactase deficient as indicated by screening test1
5. Is the volunteer apparently healthy? [No medical conditions which might affect study measurement, as judged by study physician or measured by questionnaire, and/or assessed by haematology, blood chemistry and urinalysis]
6. Is the volunteer willing to comply to study protocol during the study?
7. Is the volunteer agreeing to be informed about medically relevant personal test-results by study physician?
8. Is the volunteer willing to refrain from drinking of alcohol on and one day before the blood withdrawal?
9. Is the fasting blood glucose value of the volunteer is >3.4 and <6.1 mmol/ litre (i.e. 62-110 mg/dl)?
10. Is the Haemoglobin level within normal reference range as judged by the research physician?
11. Is the volunteer literate?

Exclusion Criteria:

1. Is the volunteer an employee of Unilever, Hindustan Lever, or Lambda Therapeutics Research?
2. Has the volunteer participated in any other biomedical study 3 months before screening visit day of this study and/or participating in any other biomedical study during the study period?
3. Does the volunteer take too much of alcohol (> 120 ml / week)?
4. Is the volunteer on a medically prescribed/slimming diet?
5. Does the volunteer work in night shifts (between 23.00 and 6.00 hrs) in the week preceding or during the study?
6. Is the volunteer using any medication including traditional medicines, vitamins, tonics which might interfere with study measurements, as judged by the PI and/or study physician?
7. Does the volunteer engage in intense exercise > 10h/week? (Intense exercise is defined as exercise which induces sweating and causes sufficient breathlessness to limit conversation)
8. Has the volunteer reported weight loss/gain > 10% of body weight in the 6 months preceding screening?
9. Has the volunteer donated any blood for 2 months prior to screening visit?
10. Does the volunteer urine analysis show any drug abuse?
11. Is the volunteer allergic to any food or cosmetics?
12. Does the volunteer smoke or consume tobacco in any form, and/or was smoking or consuming tobacco in any form for 6 months preceding the study and/or will be smoking or consuming tobacco in any form, during the study?
13. If female, is the volunteer pregnant or will she be planning pregnancy during the study period?
14. If female, is the volunteer lactating or has been lactating for 6 weeks before pre-study investigation and/or during the study period?

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2011-11-24 (Actual); Primary Completion 2012-01-06 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Post-prandial blood glucose | Positive incremental Area under the glucose versus time Curve between 0 (before) and 2 hours.
  Glucose concentration in venous plasma

SECONDARY OUTCOMES:
Breath hydrogen excretion | Fifteen minutes before (basal) and 65, 125, 185, 245, 305, 365 and 425 minutes after the ingestion of the test products
  Hydrogen gas in exhaled breath. When a subject produced 10 ppm hydrogen or more above the basal breath hydrogen level the treatment was regarded as a "positive"
Intestinal discomfort | Ten minutes before (baseline) and at 130, 250, 370 and 420 minutes after the ingestion of the test products.
  An intestinal discomfort questionnaire was administered. The questionnaire asked whether subjects had experienced 1) flatulence, 2) nausea, 3) bloating or 4) pain in the bowels. Percentage of "Yes" scores was calculated per discomfort.
Stool consistency and number of stools | 24 hours before study product intake, during 7 hour the test day and in the 17 hours after the test day (telephone interview).
  Stool consistency was evaluated by semi-quantitative Bristol scale (score between 1 = constipation and 7 = watery diarrhea).

OTHER OUTCOMES:
Post-prandial serum insulin | Total Area under the insulin versus time Curve 0-2 hours after the intake.
  Post-prandial serum insulin Area under versus time curves
Glucose in urine | Subjects were asked to empty their bladder before study product intake (-20 minutes) and again before leaving the site ( 450 minutes). In these two samples and in all additional urine samples voided while subjects were on site, glucose was analyzed
  Glucose in urine was measured using dipsticks with a detection limit of 2.28 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: David Mela, Dr., Study Director — Unilever R&D Vlaardingen (retired)
Locations (1):
- Lambda Therapeutics Research Ttd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mela DJ, Cao XZ, Dobriyal R, Fowler MI, Lin L, Joshi M, Mulder TJP, Murray PG, Peters HPF, Vermeer MA, Zhang Z. The effect of 8 plant extracts and combinations on post-prandial blood glucose and insulin responses in healthy adults: a randomized controlled trial. Nutr Metab (Lond). 2020 Jul 6;17:51. doi: 10.1186/s12986-020-00471-x. eCollection 2020. PMID 32647531